CLINICAL TRIAL: NCT05290701
Title: Evaluating Prenatal Exome Sequencing Study
Acronym: EPES
Status: Active, not recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, gwesanten, Clinical Geneticist, Leiden University Medical Center
Other Study IDs: NL77927.058.21
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Congenital Anomalies; Mendelian Disorders; Genetic Diseases, Inborn
Keywords: Prenatal diagnosis; Next Generation Sequencing; Whole Exome Sequencing; Patient perspectives; Clinical Utility
MeSH Terms: conditions — Congenital Abnormalities; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study evaluates the impact of the various outcomes of pES (definitive diagnosis, probable diagnosis and IF) on clinical decision making and on parental psychological wellbeing, compared between different analysis strategies to investigate the clinical utility, defined as the balance between potential harms and benefits.

DETAILED DESCRIPTION:
Foetal anomalies as detected on prenatal ultrasound are present in 2-3% of pregnancies. The diagnosis of a genetic syndrome as the underlying cause often has significant consequences for the prognosis and therefore also a significant impact on parental reproductive decision making. In addition to chromosomal testing, prenatal exome sequencing (pES) is increasingly being offered. Although prenatal diagnostic rates are promising, no studies report on the actual implementation of pES in routine care and thus several important knowledge gaps remain regarding clinical utility (the balance between potential harms and benefits) and the preferred analysis strategy (broad versus targeted analysis). A broad analysis has a possible higher diagnostic yield, but it is unknown whether the increased chance of finding an uncertain diagnosis and Incidental Findings outweighs this benefit when it comes to clinical decision making and parental psychological wellbeing. The central aim of this study is to address the knowledge gaps raised above, and increase clinical utility by using the obtained data to improve analysis strategies and to potentially identify new genes.

ELIGIBILITY:
Inclusion Criteria:

* At least one fetal anomaly detected in the current pregnancy, irrespective of gestational age;
* Pregnancy ongoing;
* Mother at least 18 years old and providing consent for pES;
* If father is available: father at least 18 years old and providing consent for pES.

Exclusion Criteria:

There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with one or more ultrasound findings during the current pregnancy who consent to pES, and their partner.
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of definitive diagnoses, probable diagnoses and incidental findings (IF) | 2 years

SECONDARY OUTCOMES:
Patients perspectives on probable diagnoses and incidental findings including psychological wellbeing as measured by questionnaires. | 2 years
  We will use validated scales such as the State Trait Anxiety Inventory-6, the Decisional Conflict Scale, the Decisional Regret Scale, the Intolerance of Uncertainty Scale, the Impact of Event Scale and the Pre- and Postnatal Bonding Scale.
Clinical impact of prenatal exome sequencing (pES) | 2 years
  Clinical impact will be defined as medical or surgical in utero intervention, pregnancy termination, location and mode of delivery, decisions on comfort care and neonatal policy influenced by the results of pES.
Impact of different analysis strategies on the distribution of the various outcomes of pES (definitive diagnosis, probable diagnosis and incidental findings) | 2 years
  pES data of all included pregnancies will be retrieved and re-analyzed to minimize differences in variant interpretation and to determine the impact of different analysis strategies on the percentages of various outcomes of pES (definitive diagnoses, probable diagnoses and incidental findings). Different analysis strategies will be employed: analysis of an HPO-based gene panel, analysis of an established gene panel of genes causing multiple congenital anomalies and/or intellectual disability, and analysis of all genes.

OTHER OUTCOMES:
Number of identified new disease genes | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands